CLINICAL TRIAL: NCT02660008
Title: A Randomized, Double-blind Trial of Single Doses of ZP4207 Administered s.c. to Hypoglycemic Type 1 Diabetic Patients to Describe the Pharmacokinetics and Pharmacodynamics of ZP4207 as Compared to Marketed Glucagon
Brief Title: Single Doses of ZP4207 Adm. sc to Hypoglycemic TD1 pt. to Describe the PK and PD of ZP4207 as Comp. to Marketed Glucagon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ZP4207-15126
Record Dates: First submitted 2016-01-06; First posted 2016-01-21 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Glucagon-Like Peptide 1; Glucagon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZP4207 (Experimental): ZP4207 (peptide analogue of human glucagon) Planned doses: 0.1, 0.3, 0.6, 1.0 mg s.c.
  Interventions: Drug: ZP4207
- GlucaGen (Active Comparator): GlucaGen (native glucagon) Planned doses: 0.5, 1.0 mg s.c.
  Interventions: Drug: GlucaGen

INTERVENTIONS:
Drug: ZP4207 — Parallel trial in Group 1 and cross-over trial in Groups 2-4 with single doses of ZP4207 administered s.c. to hypoglycemic Type 1 diabetic patients
  Other Names: analogue af human glucagon
  Arms: ZP4207
Drug: GlucaGen — Parallel trial in Group 1 and cross-over trial in Groups 2-4 with single doses of GlucaGen administered s.c. to hypoglycemic Type 1 diabetic patients
  Other Names: glucagon
  Arms: GlucaGen

SUMMARY:
The trial is a single-centre, randomized, double-blind, parallel trial in Group 1 and cross-over trial in Groups 2-4 with single doses of ZP4207 administered s.c. to hypoglycemic Type 1 diabetic patients to evaluate the pharmacokinetics and pharmacodynamics of ZP4207 as compared to marketed glucagon.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities (trial-related activities are any procedure that would not have been performed during normal management of the patient).
2. Male and female patients with T1D for at least one year, as defined by the American Diabetes Association.
3. Having been treated with insulin for T1D for at least 1 year.
4. Stable disease with HbA1c < 8.5%.
5. Expected stable insulin treatment during participation in trial and 3 month prior to the screening visit.
6. Age between 18 and 50 years, both inclusive.
7. Body weight between 60 and 90 kg, both inclusive.
8. Patients in good health according to age (medical history, physical examination, vital signs, ECG, lab assessments), as judged by the Investigator.

   -

Exclusion Criteria:

1. Previously treated with ZP4207.
2. Known or suspected allergy to trial product(s) or related products.
3. Previous participation (randomization) in this trial.
4. Receipt of any investigational drug within 3 months prior to screening.
5. A history or presence of cancer, or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, hematological, dermatological, venereal, neurological, psychiatric diseases, or other major diseases.
6. Clinically significant illness within 4 weeks before screening, as judged by the Investigator.
7. History of, or positive results to the screening test for Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies
8. Positive result of test for HIV antibodies.
9. Any clinically significant abnormal hematology, biochemistry or urinalysis screening tests, as judged by the Investigator.
10. Clinically significant abnormal ECG at screening as evaluated by the Investigator.
11. Donation of blood or plasma in the past month, or in excess of 500 mL within 12 weeks prior to screening.
12. A significant history of alcoholism or drug/chemical abuse, or who has a positive result in the urine drug screen, or who consumes more than 14 units of alcohol per week (one unit of alcohol equals about 250 mL of beer, 1 glass of wine, or 20 mL of spirits).
13. Habitual smoking, i.e., daily smoking or more than 7 cigarettes/week within the last 3 months prior to screening. Patients have to accept refraining from smoking while at the clinical site.
14. Patients with mental incapacity or language barriers which preclude adequate understanding or cooperation, who are unwilling to participate in the trial, or who in the opinion of the Investigator should not participate in the trial.
15. Surgery or trauma with significant blood loss within the last 2 months prior to screening.
16. Any condition interfering with trial participation or evaluation or that could be hazardous to the patient.
17. Severe hypoglycaemic events within one year prior to screening, as judged by the Investigator.
18. Significant changes in basal insulin within 3 weeks before screening, as judged by the Investigator.
19. Clinically relevant diabetic complications (macrovascular disease with symptoms or signs of coronary artery disease or peripheral vascular disease, microvascular disease with symptoms or signs of neuropathy, gastroparesis, retinopathy, nephropathy, or poor blood glucose control with polyuria, polydipsia, or weight loss), as judged by the Investigator.
20. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using highly effective contraceptive methods (highly effective contraceptive methods are considered those with a failure rate less than 1% undesired pregnancies per year including surgical sterilisation, hormonal intrauterine devices (coil), oral hormonal contraceptives, sexual abstinence or a surgically sterilised partner) or postmenopausal women being amenorrheic for less than 1 year with serum FSH level <= 40 IU/L and not using highly effective contraceptive methods during the trial and until one month after completion of the trial.
21. Male who is sexually active and not surgically sterilized who or whose partner(s) is not using highly effective contraceptive methods (highly effective contraceptive measures include surgical sterilisation, hormonal intrauterine devices [coil], oral hormonal contraceptives, each in combination with spermicide-coated condoms), or who is not willing to refrain from sexual intercourse from the first dosing until one month after last dosing in the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
PD endpoint: Plasma glucose profiles 0-360 min above baseline (Area under the effect curve 0-360 min) | During visit 2 and 3 (0-360min)
  At visit 2 and 3
PD endpoint: Time to peak plasma glucose concentration (tmax) | During visit 2 and 3 (0-360min)
  At visit 2 and 3
PK endpoint: Plasma ZP4207 and glucagon profiles 0-360 min | During visit 2 and 3 (0-360min)
  At visit 2 and 3
PK endpoint: Peak plasma concentration (Cmax) | During visit 2 and 3 (0-360min)
  At visit 2 and 3
PK endpoint: Time to peak plasma concentration (tCmax) | During visit 2 and 3 (0-360min)
  At visit 2 and 3

SECONDARY OUTCOMES:
PD endpoints: Percentage of patients achieving a plasma glucose concentration ≥70 mg/dL within 30 minutes after treatment | During visit 2 and 3 (0-30min)
  At visit 2 and 3
PD endpoints: Time to plasma glucose concentration of ≥70 mg/dL | During visit 2 and 3 (0-360min)
  At visit 2 and 3
PD endpoints: Percentage of patients achieving a plasma glucose increase of ≥20 mg/dL within 30 minutes after treatment | During visit 2 and 3 (0-30min)
  At visit 2 and 3,
PD endpoints: Time to plasma glucose increase of ≥20 mg/dL | During visit 2 and 3 (0-360min)
  At visit 2 and 3,
PK endpoints: Baseline adjusted glucagon profiles 0-360 min | During visit 2 and 3 (0-360min)
  At visit 2 and 3,
PK endpoints: AUC0-inf for plasma ZP4207 concentration | During visit 2 and 3 (0-360min)
  At visit 2 and 3, Area under the plasma curve from 0 to infinity
Exploratory endpoint: Insulin concentrations | During visit 2 and 3 (0-360min)
  At visit 2 and 3, insulin concentrations in serum
Exploratory endpoint: Changes in hypoglycaemic symptom scores from 0-30 minutes | During visit 2 and 3 (0-30min)
  At visit 2 and 3
Safety and Tolerability: Number of participants with adverse events | Through study completion (up to 63 days)
  Number of participants with adverse events
Safety and Tolerability: Changes or findings from baseline in physical examination | Through study completion (up to 63 days)
  An examination of the following body systems will be performed:
  * Head, ears, eyes, nose, throat (HEENT), incl. thyroid gland
  * Heart, lung, chest
  * Abdomen
  * Skin and mucosae
  * Musculoskeletal system
  * Nervous system
  * Lymph node
  * Other findings
Safety and Tolerability: Changes or findings from baseline (normal ranges) in clinical safety laboratory parameters | Through study completion (up to 63 days)
  Haematology biochemistry, and urinalysis
Safety and Tolerability: Changes or findings from baseline in vital signs | Through study completion (up to 63 days)
  systolic/diastolic blood pressure (mmHg) and heart rate (beats per minute), body temperature (°C), respiratory frequency (RF/min)
Safety and Tolerability: Changes or findings from baseline in ECG | Through study completion (up to 63 days)
  Heart rate, PQ, QRS, QT, QTcB
Safety and Tolerability: Local tolerability of injection site | Through study completion (up to 63 days)
  Findings in local tolerability by means of the following assessments.
  * spontaneous pain
  * pain on palpation
  * itching
  * redness
  * oedema
  * induration/infiltration
  * other
Safety and Tolerability: Immunogenicity (Ant-Drug Antibody sampling) | Through study completion (up to 63 days)
  Antidrug antibodies incidences

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

REFERENCES:
- [Derived] Hovelmann U, Bysted BV, Mouritzen U, Macchi F, Lamers D, Kronshage B, Moller DV, Heise T. Pharmacokinetic and Pharmacodynamic Characteristics of Dasiglucagon, a Novel Soluble and Stable Glucagon Analog. Diabetes Care. 2018 Mar;41(3):531-537. doi: 10.2337/dc17-1402. Epub 2017 Dec 22. PMID 29273578